CLINICAL TRIAL: NCT03158181
Title: Improvement of Intraoperative Behavior of Staff to Prevent Postoperative Complications
Acronym: ARIBO2
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0076
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Complications
Keywords: Behavior; Operational block; Monitoring; Social Sciences ; New technologies
MeSH Terms: conditions — Postoperative Complications; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional study — None intervention will be conduct on patient. Only the operating room will be randomized to have an intervention or not (Bundle of measure for optimizing the discipline of personnel in the operating room)

SUMMARY:
The aim of this interventional study is to optimize the movements and discipline of surgical staff in order to improve the quality of care, the safety of the patient in the surgery and to prevent the postoperative complications in the broad sense and in particular the infection of the surgical site. The intervention will be carried out using tools of new technologies allowing the monitoring of the movements and the sound level associated with techniques of behavior change inspired by those used in the human and social sciences.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient agreeing to participate in the study
* Patient who will benefit from orthopedic surgery for hip or knee arthroplasty with prosthesis placement

Non-Inclusion Criteria:

* Patient with previous history of surgical site infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients receiving hip and knee prosthetic prosthetic orthopedic surgery on a scheduled and emergency first-line basis.
  This choice is due to the following reasons:
  This specialty requires a cutaneous approach, All these gestures are Altemeier class I or own surgery, These are frequent surgeries, the most frequent in orthopedics They are reproducible acts allowing the comparison from one center to another.
Sampling Method: Non-Probability Sample
Enrollment: 20959 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of any major postoperative complications | Until 30 days after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel BIRGAND, Dr, Principal Investigator — Nantes University Hopital
Locations (16):
- France (16):
  - Angers University Hospital, Angers
  - Vendée Hospital, La Roche-sur-Yon
  - Pré surgical clinic, Le Mans
  - Le Mans Hospital, Le Mans
  - Nantes University Hospital, Nantes
  - H.P. Confluent, Nantes
  - Hôpital Lariboisière, Paris
  - IMM, Paris
  - Hôpital Beaujon, Paris
  - Rennes University Hospital, Rennes
  - Saint Grégoire private hospital, Saint-Grégoire
  - Sante Atlantique, Saint-Herblain
  - Saint-Nazaire Hospital, Saint-Nazaire
  - Tours University Hospital, Tours
  - Saint-Léonard Clinic, Trélazé
  - Vannes Hospital, Vannes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birgand G, Haudebourg T, Grammatico-Guillon L, Ferrand L, Moret L, Gouin F, Mauduit N, Leux C, Le Manach Y, Lepelletier D, Tavernier E, Lucet JC, Giraudeau B. Improvement in staff behavior during surgical procedures to prevent post-operative complications (ARIBO2): study protocol for a cluster randomised trial. Trials. 2019 May 20;20(1):275. doi: 10.1186/s13063-019-3370-z. PMID 31109343